CLINICAL TRIAL: NCT03840980
Title: The Alberta BLOOM Preterm Neonate Study: The Impact of Perinatal Factors on the Microbiome, Immunobiome, and Metabolome of Preterm Neonates
Brief Title: The Alberta BLOOM Preterm Neonate Study
Acronym: BLOOM-PTN
Status: Terminated | Type: Observational
Why Stopped: The BLOOM-PTN study has evolved into the ongoing BLOOM-PCS study (REB20-1442)
Sponsor: University of Calgary (Other)
Collaborators: Alberta Economic Development and Trade (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: REB17-1877
Record Dates: First submitted 2018-12-19; First posted 2019-02-15 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Infant, Premature; Infants, Extremely Premature; Microbiota; Gastrointestinal Microbiome
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, Stool, Breast Milk, Whole Blood, Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational clinical cohort study involving 100 mothers and their very preterm infants born at less than 32 weeks gestation. The purpose of this study is to gain a thorough understanding of the microbiome (the collection of microbes in a biological site) establishment in very preterm infants. The study will also examine the perinatal factors associated with the pattern of microbiome development, the metabolome and immune development of this population in the first months of life.

All participants will be recruited from the Neonatal Intensive Care Unit (NICU) at Foothills Medical Centre (FMC) in Calgary, Alberta, Canada.

Premature birth (birth before 37 weeks of pregnancy) occurs in about one in ten pregnancies each year. Babies that are born after less than 32 weeks of pregnancy are considered to be very premature babies. When babies are born very prematurely their gut is not as developed. One important factor in gut health is the large community of microbes (tiny living things such as bacteria) that live on the human body called the microbiome. Recent studies have shown that premature babies are more likely to have changes in their gut microbiome that are associated with health issues. However, sciences has not yet discovered what specific microbiome features are involved in development of premature babies. Therefore, this study examines the impact of very premature birth on the premature baby's microbiome.

The kind of microbes that make up the microbiome in the gut in the first months of life have a major impact on the microbiome that will form during childhood. There are many environmental factors during pregnancy, birth and in first months of life that can impact the microbiome development. These factors include diet, exposure to antibiotics, surgical procedures, and birth mode. This study will investigate how these factors influence the types of early microbes present in preterm infants.

The hypothesis of the study is that specific microbial patterns, trajectories and/or metabolites will be significantly associated with single or a combination of perinatal maternal and/or infant factors.

The primary objective of the study is to learn more about the development of the microbiome in very premature babies in the first months of their life. To do this, participating baby's stool and urine samples will be studied.

A secondary objective of the study is to find out how environmental factors impact the development of the microbiome and the health of preterm infants. In order to do this, maternal microbiome samples will be studied and information regarding maternal health, nutrition and environment during pregnancy will be collected. As well, information about the birth and health of participating preterm neonates will be collected.

ELIGIBILITY:
Infant Inclusion Criteria:

1. Born within previous 72 hours;
2. Born at ≤ 31 weeks + 6 days gestation (31 6/7 weeks);
3. Expected to survive more than 1 week;
4. Admitted into the Neonatal Intensive Care Unit at Foothills Medical Centre, Calgary, Alberta;
5. Have no major congenital or chromosomal anomalies.

Mother Inclusion Criteria

1. Provide a signed and dated informed consent form;
2. Able to speak and understand English;
3. 16 years of age or older (if 16 or 17 years of age, must be documented in the patient's health record to be a mature minor / competent to provide consent);
4. Willing to comply with all study procedures and be available for the duration of the study;
5. Reside within the Calgary Metropolitan Region.

Infant Exclusion Criteria

1) Has congenital gastrointestinal anomalies or has a history of gastrointestinal surgery.

Mother Exclusion Criteria

1. Not the legal guardian of the baby or
2. In a legal guardianship dispute.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Due to the observational nature of this study and the need to understand early microbiome assembly in all very preterm babies, regardless of the pregnancy complication that led to their premature birth, this study aims to recruit most very preterm neonates that are expected to survive more than one week. Neonates with congenital gastrointestinal anomalies or that have a history of gastrointestinal surgery, will be excluded as these conditions severely affect the microbiome; however the microbiome will not have contributed to the development of these conditions. Participants must reside in the Calgary Metropolitan Region in order to ensure that they can be followed for study participation if transferred to a level II NICU or discharged to home. Only mothers able to legally consent to study participation for themselves and their neonate are eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Microbiome | First 5-6 months of life
  Fecal microbial diversity and the relative abundance of bacterial and eukaryotic taxa, as assessed by polymerase chain reaction of the 16S and ITS2 gene and functional analysis on 16S taxonomic surveys for all participants from birth through to 60 days of age.
Microbiome Assembly | First 5-6 months of life
  Changes in fecal microbial diversity and microbial population structures from birth through to 60 days of age for all participants as assessed by shotgun metagenomics.
Metabolome | First 5-6 months of life
  Human and microbial metabolites as assessed by untargeted metabolomics, ultra performance liquid chromatography ultrahigh-resolution Fourier transform (FT) combined with mass spectrometry to identify human and microbial metabolites for all participants from birth through to 60 days of age.
Immunobiome | First 5-6 months of life
  Immune analysis of cytokines and chemokines as assessed by mesoscale system for participants with suspected infection such as NEC or neonatal sepsis in the 60 days of study participation.

SECONDARY OUTCOMES:
Perinatal factors and microbiome, metabolome and immunobiome. | first 5-6 months of life
  Association between perinatal factors (environment, nutrition, pharmacological exposure), preterm delivery and the patterns of microbiome, metabolome and immunobiome development as assessed by metagenomics, metabolomics and mesoscale analysis for all participants in the first 60 days of life.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claire Arrieta, PhD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- See also: Alberta BLOOM Study Website — http://albertabloom.ca/